CLINICAL TRIAL: NCT04160208
Title: DNA Damage and Subfertility in Males - Impact on Assisted Reproductive Treatment Outcome
Brief Title: DNA Damage and Subfertility in Males - Impact on ART Outcome
Acronym: ReproDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Other Study IDs: DFI2019Skivecohort
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Infertility
Keywords: male infertility; DNA fragmentation Index; DFI
MeSH Terms: conditions — Infertility; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- IUI - Insemination: Males of couples undergoing their first IUI treatment
- IVF - In vitro fertilisation: Males of couples undergoing their first IVF treatment. Including males of couples who have had previous IUI treatments.
- ICSI - Micro Insemination: Males of couples undergoing their first ICSI treatment. Including males of couples who have had previous IUI treatments.

SUMMARY:
A obvational prospective cohort study of men undergoing IUI, IVF and ICSI treatment in Denmark. The aim is to asses the impact of sperm DNA damage, measured as DNA fragmentation index (DFI), on reproductive outcomes after assisted reproductive technology (ART).

ELIGIBILITY:
Inclusion Criteria:

* First cycle treatment

Exclusion Criteria:

* TESA/PESA, more than one cycle

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males of couples attending Skive fertility Clinic
Sampling Method: Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of particpants achieving live birth | week 23-42 of pregnancy
  Birth of a living child after week 23. Registered through self-reported schemes sent to the clinic.

SECONDARY OUTCOMES:
Number of participants with clinical pregnancy | week 7-8 of pregnancy
  Measurement of heart beat by ultrasound scan
Number of participants with biochemical pregnancy | Day 14-17 of pregnancy
  Increase in serum hCG levels
Cumulative live birth rate | 9-24 months after inclusion
  Live births originating from one controlled stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Skive Regional Hospital, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No